CLINICAL TRIAL: NCT00089531
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of a 6-Plasmid Multiclade HIV-1 DNA Vaccine, VRC-HIVDNA016-00-VP, in Uninfected Adult Volunteers
Brief Title: Candidate HIV Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040254; 04-I-0254
Record Dates: First submitted 2004-08-05; First posted 2004-08-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-01-15

CONDITIONS: HIV Infections
Keywords: Healthy; Virus; T-Cells; HIV-Negative; Immunity; Healthy Volunteer; HV; HIV Preventive Vaccine; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Virus Diseases

INTERVENTIONS:
Drug: VRC-HIVDNA016-00-VP

SUMMARY:
This study will evaluate whether an experimental vaccine intended to prevent HIV infection is safe and whether it causes any side effects. It will also examine whether the vaccine, called VRC-HIVDNA016-00-VP, causes an immune response, and will monitor participants for the social impact of being in an HIV vaccine study. VRC-HIVDNA016-00-VP contains synthetic DNA that codes for parts of four HIV proteins. It also contains a "promoter" piece of DNA that is needed to start protein production. The promoter DNA is also synthetic and is like the promoter in another virus called cytomegalovirus (CMV). The vaccine contains no live HIV virus or CMV and cannot cause either of these illnesses.

Healthy volunteers between 18 and 44 years old who are HIV-negative may be eligible for this 32-week study. Candidates are screened with a medical history, physical examination, and blood and urine tests.

Participants receive three injections of the experimental vaccine approximately 28 days apart. The injections are given with a system called the Biojector 2000 that delivers the vaccine through the skin into the muscle without the use of a needle. Subjects are observed for side effects for at least 30 minutes after each vaccination and are required to telephone the clinic staff 1 to 2 days after the injection to report how they are doing. In addition, they are given a diary card to take home, on which they record their temperature and any symptoms daily for five days.

Participants return to the clinic two weeks after each injection. They return the completed diary card and are checked for any health changes or problems since the last visit. They are asked how they are feeling and what medications, if any, they have taken. Blood and urine samples are collected. Some subjects may be asked to have laboratory tests between regular visits if needed to evaluate a change in health. Participants are also asked about any social effects they may have experienced as a result of their participation in the study.

DETAILED DESCRIPTION:
Study Design: This is a Phase I open label study to evaluate safety, tolerability, and immune response of a 6-plasmid multiclade HIV-1 DNA vaccine, VRC-HIVDNA016-00-VP. The hypothesis is that this regimen will be safe for human administration and elicit immune responses to HIV-1 clade B Gag, Pol and Nef proteins, as well as clades A, B and C Env proteins. The primary objective is to evaluate the safety and tolerability in humans of the investigational vaccine and secondary objectives are to evaluate the immunogenicity of the vaccine as measured by intracellular cytokine staining (ICS) in the 4 weeks after the second or third dose of vaccine and the social impact of participating in an HIV-1 vaccine trial.

Product Description: VRC-HIVDNA016-00-VP is composed of 6 closed, circular DNA plasmids that are each 16.67 percent (by weight) of the vaccine. Each of the 6 plasmids in this vaccine expresses a single gene product. Plasmids VRC 4401, VRC 4409 and VRC 4404 are designed to express clade B HIV-1 Gag, Pol and Nef, respectively. VRC 5736, VRC 5737, and VRC 5738 are designed to express HIV-1 Env glycoprotein from clade A, clade B, and clade C, respectively. Vaccine vials will be supplied at 4 mg/mL. Each DNA vaccination will be 1 mL of vaccine administered intramuscularly (in deltoid muscle) using the Biojector 2000 Needle-Free Injection Management System.

Subjects: Healthy adult volunteers (18 to 44 years old) will be enrolled.

Study Plan: Fifteen volunteers will be enrolled, as shown in the schema:

Name of Vaccine: VRC-HIVDNA016-00-VP

Number of Subjects: 15

Vaccine Injection Schedule: (at least 21 days between injections)

Day 0: 4 mg

Day 28 plus or minus 7: 4 mg

Day 56 plus or minus 7: 4 mg

Study Duration: 32 weeks clinical follow-up for each participant.

Study Endpoints: The primary endpoint is safety of the regimen; secondary endpoints are

cellular immune responses as measured by ICS within the first 4 weeks after the second and

third doses and social impact at Week 32. Exploratory analyses will include HIV-specific

antibody assays, ICS or other immunological assays at intervals between Day 0 and Week 32.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must meet all of the following criteria:

18 to 44 years old.

Available for clinical follow-up through Week 32 of the study.

Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.

Complete an Assessment of Understanding prior to enrollment and verbalize understanding of all questions answered incorrectly.

Able and willing to complete the informed consent process.

Willing to receive HIV test results and willing to abide by NIH guidelines for partner notification of positive HIV results.

Willing to donate blood for sample storage to be used for future research.

Willing to discuss HIV infection risks and amenable to risk reduction counseling.

In good general health without clinically significant medical history and has satisfactorily completed screening.

Physical examination and laboratory results without clinically significant findings within the 28 days prior to enrollment.

Laboratory Criteria within 28 days prior to enrollment:

Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to 13.5 g/dL for men.

WBC equal to 3,300-12,000 cells/mm(3).

Differential either within institutional normal range or accompanied by site physician approval.

Total lymphocyte count greater than or equal to 800 cells/mm(3).

Platelets equal 125,000 - 550,000/mm(3).

ALT (SGPT) less than or equal to 1.25 x upper limit of normal.

Serum creatinine less than or equal to upper limit of normal.

Normal urinalysis defined as negative glucose, negative or trace protein, and negative or trace hemoglobin (blood).

Negative FDA-approved HIV blood test.

Negative Hepatitis B surface antigen.

Negative anti-HCV.

Female Specific Criteria:

Negative beta-HCG pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.

A female participant must meet any of the following criteria:

No reproductive potential because of menopause (one year without menses) or because of a hysterectomy, bilateral oophorectomy, or tubal ligation,

OR

Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and through Week 32 of the study,

OR

Participant agrees to consistently practice contraception at least 21 days prior to enrollment and through Week 32 of the study by one of the following methods:

Condoms, male or female, with or without a spermicide;

Diaphragm or cervical cap with spermicide;

Intrauterine device;

Contraceptive pills or patch, Norplant, Depo-Provera or other FDA-approved contraceptive method;

Male partner has previously undergone a vasectomy for which there is documentation.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

Women:

Woman who is breast-feeding or planning to become pregnant during the 32 weeks of study participation.

Volunteer has received any of the following substances:

HIV vaccines in a prior clinical trial;

Immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis);

Blood products within 120 days prior to HIV screening;

Immunoglobulin within 60 days prior to HIV screening;

Investigational research agents within 30 days prior to initial study vaccine administration;

Live attenuated vaccines within 30 days prior to initial study vaccine administration.

Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days of study vaccine administration;

Current anti-TB prophylaxis or therapy.

Volunteer has a history of any of the following clinically significant conditions:

Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain.

Autoimmune disease or immunodeficiency.

Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.

Diabetes mellitus (type I or II), with the exception of gestational diabetes.

History of thyroidectomy or thyroid disease that required medication within the past 12 months.

Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years.

Hypertension that is not well controlled by medication or is more than 150/100 at enrollment.

Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.

Syphilis infection that is active or a positive serology due to a syphilis infection treated less than six months ago.

Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.

Seizure disorder other than:

1. febrile seizures under the age of two,
2. seizures secondary to alcohol withdrawal more than 3 years ago, or
3. a singular seizure not requiring treatment within the last 3 years.

Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.

Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years; disorder requiring lithium; or suicidal ideation occurring within five years prior to enrollment.

Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15
Dates: Start 2004-08-02; Study Completion 2008-01-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Casimiro DR, Chen L, Fu TM, Evans RK, Caulfield MJ, Davies ME, Tang A, Chen M, Huang L, Harris V, Freed DC, Wilson KA, Dubey S, Zhu DM, Nawrocki D, Mach H, Troutman R, Isopi L, Williams D, Hurni W, Xu Z, Smith JG, Wang S, Liu X, Guan L, Long R, Trigona W, Heidecker GJ, Perry HC, Persaud N, Toner TJ, Su Q, Liang X, Youil R, Chastain M, Bett AJ, Volkin DB, Emini EA, Shiver JW. Comparative immunogenicity in rhesus monkeys of DNA plasmid, recombinant vaccinia virus, and replication-defective adenovirus vectors expressing a human immunodeficiency virus type 1 gag gene. J Virol. 2003 Jun;77(11):6305-13. doi: 10.1128/jvi.77.11.6305-6313.2003. PMID 12743287